CLINICAL TRIAL: NCT06839365
Title: Breaking the Silence: A Cross-Sectional Study on Barriers to Mental Health Help-Seeking Among Egyptian Medical Students
Brief Title: A Cross-Sectional Study on Barriers to Mental Health Help-Seeking Among Egyptian Medical Students
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Saad Elsaeidy, Dr., Benha University
Other Study IDs: RC 5-3-2022
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Mental Health Conditions
Keywords: Mental health, help-seeking, Students, Family, Al-Azhar, Suicide.
MeSH Terms: conditions — Psychological Well-Being; Suicide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Egyptian medical students: Young adult medical students aged 18 to 25 in the different Egyptian faculties of medicine and from different medical class years were eligible to participate. During the recruitment of the participants, we used convenience and snowball sampling techniques.

SUMMARY:
High levels of mental distress were reported among medical students; however, only a small portion decided to seek help. This study aims to identify the most diagnosed mental disorders among medical students in Egypt, recognising their family attitudes and the major barriers that deter them from seeking help. This is a cross-sectional study conducted on Egyptian medical students.

DETAILED DESCRIPTION:
Study design A multicenter cross-sectional study across Egypt was conducted among Egyptian medical students via different social media platforms of the Egyptian faculties of medicine.

Study population Data collection Young adult medical students aged 18 to 25 in the different Egyptian faculties of medicine and from different medical class years were eligible to participate. During the recruitment of the participants, we used convenience and snowball sampling techniques. The online survey and data collection took place from April to June 2022.

Sample Size Calculation The sample size was calculated using the equation (n = [Z2 × P (1-P)] ÷ e2) [14] Under a 95% Confidence level (Z=1.96), 50% response distribution (P=0.5) and confidence interval (e=3), a sample of 1067 participants were required.

Measurements The participants were presented with an online and self-administered questionnaire including 27-item barriers mentioned in the 30-item Barriers to Access to Care Evaluation (BACE) scale [15]. Each questionnaire consisted of 4 sections: the first was assessing the sociodemographic characteristics of the participants. The second was assessing the presence of previously diagnosed mental disorders. The third was the 27-item BACE survey including 9 items for the stigma, 10 for the altitudinal barriers, 6 for instrumental barriers, and 2 work-related items preceded by a question if the student works or not; the 2 items of work were reallocated from the stigma and instrumental sections, based on the assumption that only small portion of the medical students has an occupation. The last segment was family-related yes-or-no questions assessing the family attitude towards mental health (by asking if they know mental health's importance if they recognize it as important as physical health and their support in the presence of mental health problems) and the presence or absence of previous familial suicidal attempts.

Data analysis Data were analysed using SPSS version 25. The internal consistency of the survey was determined using Cronbach's α. The internal consistency of the overall 27-item scale (stigma, attitudinal, instrumental, and working-beside-education barriers) was of good reliability (α = 0.904). We used the frequency and percentage to summarise the categorical data but mean and standard division to summarise the total effect of each domain. The Chi-square test, Fisher's exact test, and odds ratio (OR) were carried out on categorical data. The three-point Likert scale was used to determine whether the barrier is considered not a barrier, a minor barrier, or a major barrier using Likert intervals (0, 0.67, 1.34, 2). A P-value of ≤ 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

Young adult medical students aged 18 to 25 in the different Egyptian faculties of medicine and from different medical class years were eligible to participate

Exclusion Criteria:

not Young adult medical students aged 18 to 25 in the different Egyptian faculties of medicine and from different medical class years were eligible to participate

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adult medical students aged 18 to 25 in the different Egyptian faculties of medicine and from different medical class years were eligible to participate
Sampling Method: Probability Sample
Enrollment: 1037 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Barriers to Access to Care Evaluation (BACE) scale | data collection took place from April to June 2022
  The participants were presented with an online and self-administered questionnaire including 27-item barriers mentioned in the 30-item Barriers to Access to Care Evaluation (BACE) scale

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Benha University, Banhā, Egypt
  - Benha University, Banhā

IPD SHARING:
Plan to Share IPD: No